CLINICAL TRIAL: NCT05828394
Title: Palate Wound Healing and Pain Perception of De-epthelized Ctg vs Sub-epithelial Ctg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Gonzalo Blasi, Principal Investigator Gonzalo Blasi, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PER-ECL-2021-07
Record Dates: First submitted 2023-02-16; First posted 2023-04-25 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Palate; Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Depithelised Free Gingival Graft, DFGG (Experimental): The group assignment was communicated through a sealed envelope that was opened just prior to the surgery. The subjects will undergo to a harvesting procedure of a palatal graft using DFGG technique described as following: two horizontal and two vertical incisions will be traced with a 15C blade to delimit the area to be grafted. Along the coronal horizontal incision, the blade will be oriented almost perpendicular to the bone plate and once an adequate soft tissue thickness was obtained, it will be rotated in order to be almost parallel to the superficial surface. The thickness of the graft will be maintained uniform while proceeding apically with the blade. Once the graft is separated, the adipose and glandular tissue as well as the epithelium will be removed extra orally with a new blade. Finally the palate will be sutured with 5-0 monofilament suture and collagen sponges. In this group the palate is suppose to have a secondary intention healing.
  Interventions: Procedure: DFGG
- Subepithelial Connective Tissue Graft, SCTG (Experimental): The group assignment was communicated through a sealed envelope that was opened just prior to the surgery. The subjects will undergo to a harvesting procedure of a palatal graft using SCTG technique described as following: one deep horizontal incision parallel to the gingival margin will be traced at 1.5 mm apical to the gingival margin of the adjacent teeth, according to the palatal pocket depth of the teeth. A deeper incision parallel and deeper to the initial one will be performed. The primary flap will be elevated split-thickness. The horizontal incision will be made almost perpendicular to the underlying bone. Once an adequate soft tissue thickness is obtained, the blade will be rotated in order to be almost parallel to the external surface. The thickness of the graft will be maintained uniform. Finally the palate will be sutured with 5-0 monofilament suture and collagen sponges.In this group the palate is suppose to have a primary intention healing.
  Interventions: Procedure: SCTG

INTERVENTIONS:
Procedure: DFGG — Depithelised free gingival graft harvesting technique
  Arms: Depithelised Free Gingival Graft, DFGG
Procedure: SCTG — Subepithelial connective tissue graft harvesting technique
  Arms: Subepithelial Connective Tissue Graft, SCTG

SUMMARY:
A single blinded randomized clinical trial was designed to evaluate the influence of palatal harvesting technique on post-operatory patient pain perception. The participants will be selected between subjects in need of at least one mucogingival procedure involving the harvesting of a connective tissue graft and then randomly allocated in the following groups. Two harvesting techniques were chosen to be compared: de-epithelialized free gingival graft (DFGG) and subepithelial connective tissue graft (SCTG).

DETAILED DESCRIPTION:
To evaluate the postoperative pain, patients were instructed to complete a 100-mm VAS and classify the level of pain experienced on the palatal site from 0 to 10, with 10 being the worst pain ever experience. Analgesics intake (AI): Post-operative pain was indirectly evaluated on the basis of the mean mg consumption of analgesics (ibuprofene). Post operative complications (PC): To evaluate the excessive bleeding., patients were instructed to complete a 100-mm VAS and classify the level of bleeding experienced on the palatal site from 0 to 10. Dimensions of the needed graft (GD0): (x0=length, y0=height, z0=thickness) it will be measured once prepared the recipient site.

Dimensions of the harvested graft (GD1): (x1=length, y1=height, z1=thickness) it will be measured with a calliper calibrated in mm just after the harvesting. Surgical time (T): time required from harvesting the graft till the suture of the donor site. Intra surgical complications (IP): perforations of the palatal flap (in the case of the SCTG) and arterial bleeding will be registered and counted as intra-surgical complications. The following parameters will be calculated:

Palatal volume changes (V changes): Volumetric differences between the intraoral scans of baseline and at every following recall will be assessed with the aim of software (Geomagic by 3d systems). Superimposing the STL files using the teeth as fixed reference points will allow to measure differences in volume changes. Graft dimensions accuracy (GDA): It will be assessed comparing GD0, the needed dimensions of the graft (x0=length, y0= height, z0= thickness) with GD1, the actual dimensions of the harvested graft (x1=length, y1= height, z1= thickness). Mean baseline thickness of the palatal soft tissues (mT0): It will be measured superimposing the cbct with the intraoral scan at baseline. The measurements will be performed using a implant planning software. Mean final thickness of the palatal soft tissues (mT1): It will be measured superimposing the cbct with the intraoral scan at 12 weeks. The measurements will be performed using a implant planning.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 18 years
* Systemically healthy
* Healthy periodontium or demonstrating stable periodontal condition following conventional periodontal therapy
* Full mouth plaque score (FMPS) and full mouth bleeding score (FMBS) of < 15%
* Non-smokers or smokers of ≤ 10 cigarettes per day
* Indication of mucogingival surgery in teeth and/or implants.

Exclusion Criteria:

* Smokers ≥ 10 cigarettes per day
* General contraindications for surgery
* Medications known to affect the gingiva or interfere with wound healing
* Pregnancy
* Benzodiazepines and/or analgesics intake
* Patients nos systemically healthy or uncontrolled (i.e: Diabetes, inmunosuppresed)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Volumetric changes during wound healing | At baseline and at 1, 2, 3, 4, 6, 8, 10 and 12 weeks after the intervention
  Volumetric differences of the harvested site between baseline (prior to the intervention) and every following recall will be assessed. Intraoral scans will be registered at baseline and at 1, 2, 3, 4, 6, 8, 10 and 12 weeks after the intervention during healing. The results will be elaborated superimposing the STL files registered at very time points using Geomagic software (3d systems). The software will output a descriptive statistics: mean volumetric difference, Minimum, Maximum, Variance.

SECONDARY OUTCOMES:
Patients pain perception | At baseline and at 1, 2, 3, 4, 6, 8, 10 and 12 weeks after the intervention
  To evaluate the postoperative pain, patients were instructed to to fill a questionnaire at every time point. The questionnaire consisted of a 100-mm Visual Analog Scale (VAS) describing the level of pain experienced on the palatal site from 0 to 10, with 10 being the worst pain ever experience, and 0 no pain.
Analgesics Intake | At baseline and at 1, 2, 3, 4, 6, 8, 10 and 12 weeks after the intervention
  Post-operative pain was indirectly evaluated on the basis of the mean mg (milligrams) consumption of analgesics (ibuprofene).
Histological Analysis | During surgery
  Tissue samples (1 × 1 × 5 mm) harvested will be fixed in buffered 4% formaldehyde overnight. After a routine preparation for paraffin embedment including tissue immersion in a series of alcohol baths at different concentrations, the specimens will be sectioned (3 μm) with a Rotatory Microtome CUT4062 and stained with hematoxylin-eosin. The obtained sections will be examined using a Leica DMR microscope and photographed with a Leica DFC 320 digital camera. The histo-morphometrical analysis will be conducted using an image processing software with the assessment of total area of the sample (TAS), area of epithelium (AE), area of lamina propria (ALP), area of submucosa (ASM), and the average epithelium thickness (ET) measured in three different locations in each sample.
Immunohistoquemical Analysis of S100 protein | During surgery
  S100 protein is characteristic of nervous tissues cells. This analysis aim to compare the subjective pain perception of other outcomes with the quantity of nervous cells found in the graft. Sections will be cut, dewaxed and rehydrated. Antibodies, along with their dilutions and sources. For antigen retrieval, heat treatments will be applied (95°C, 8 min in cell conditioning solution 1 for Glut1, calretinin and S100, and cell conditioning solution 2 for Map2) prior to the primary antibody reactions. A Tris-based buffer solution (pH 7.6 ± 0.2) was used. After UV inhibition, primary antibody reactions will be performed, in addition to counterstaining with haematoxylin. Neurone specific enolase staining will be performed. The immuno-histoquemical analysis will be conducted using an image processing software with the assessment of total area of the sample in order to count ganglia and neurons in an area of up to five high power fields in relation to it.
Graft dimension accuracy | During surgery
  Graft dimensions accuracy (GDA): It will be assessed comparing GD0, the needed dimensions of the graft (x0=length, y0= height, z0= thickness), registered in advanced, with GD1, the actual dimensions of the harvested graft (x1=length, y1= height, z1= thickness).
post-srugical pain | At baseline and at 1, 2, 3, 4, 6, 8, 10 and 12 weeks after the intervention
  the following questions, both assessed at every recall. (1) Did you take any more painkillers due to the palatal pain since the procedure was completed? (2) If necessary, would you repeat the palatal harvesting procedure? (3) Did you have any unexpected post-operative incidence? Whenever the patient stopped to take analgesics the measurement of this outcome will be interrupted. Being answered by yes or no.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Universidad Internacional de Catalunya, Sant Cugat del Vallès, Barcelona
  - International University of Catalunya, Barcelona

IPD SHARING:
Plan to Share IPD: No